CLINICAL TRIAL: NCT03702426
Title: Comparison of the Efficacy of Granulocyte - Macrophage Colony Stimulating Factor (GM-CSF) and Norfloxacin in Secondary Prophylaxis for Spontaneous Bacterial Peritonitis - A Randomised Controlled Trial
Brief Title: Comparison of the Efficacy of Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) and Norfloxacin in Secondary Prophylaxis for Spontaneous Bacterial Peritonitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-SBP-01
Record Dates: First submitted 2018-09-24; First posted 2018-10-11 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Spontaneous Bacterial Peritonitis
MeSH Terms: interventions — Norfloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Norfloxacin with GM-CSF (Experimental): Oral Norfloxacin 400mg daily and GM-CSF (Granulocyte-Macrophage colony-stimulating factor) in a dose of 1.5mcg/kg over 4 hour infusion every 15 days will be given in Group B
  Interventions: Drug: GMCSF; Drug: Norfloxacin
- Norfloxacin (Active Comparator): Patients who fulfil the inclusion criteria will receive oral norfloxacin 400 mg daily as secondary prophylaxis for SBP in Group A.
  Interventions: Drug: Norfloxacin

INTERVENTIONS:
Drug: GMCSF — GMCSF 1.5mcg/Kg
  Arms: Norfloxacin with GM-CSF
Drug: Norfloxacin — Tablet Norfloxacin 400 mg

SUMMARY:
-Consecutive patients of decompensated cirrhosis of any etiology, presenting to the Institute of Liver and Biliary Sciences hospital with spontaneous bacterial peritonitis will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 70years
* Patients of decompensated liver cirrhosis who present with spontaneous bacterial peritonitis (Presence of more than 250 neutrophils per cc of ascitic fluid, in the absence of a surgical abdomen, in the presence of decompensated cirrhosis and portal hypertension) that has responded to standard medical care.

Exclusion Criteria:

* Allergic to quinolones
* Advanced HCC (Hepatocellular Carcinoma)
* Post liver transplant
* HIV (Human Immunodeficiency Virus) positive patients
* Patients on immunosuppressive therapy
* Pregnancy
* Acute Liver Failure
* History of hematological malignancy or bone marrow transplantation
* No informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Spontaneous Bacterial Peritonitis on secondary prophylaxis in both groups | 6 Month
  Spontaneous Bacterial Peritonitis is defined as Polymorphonuclear count > 250 in ascitic fluid

SECONDARY OUTCOMES:
Survival in both groups after development of SBP (Spontaneous Bacterial Peritonitis ). | 4 weeks
  Spontaneous Bacterial Peritonitis is defined as Polymorphonuclear count > 250 in ascitic fluid.
Survival in both groups after development of SBP (Spontaneous Bacterial Peritonitis ). | 12 weeks
  Spontaneous Bacterial Peritonitis is defined as Polymorphonuclear count > 250 in ascitic fluid.
Survival in both groups after development of SBP (Spontaneous Bacterial Peritonitis ). | 24 weeks
  Spontaneous Bacterial Peritonitis is defined as Polymorphonuclear count > 250 in ascitic fluid.
Survival in both groups after development of SBP (Spontaneous Bacterial Peritonitis ). | 48 weeks
  Spontaneous Bacterial Peritonitis is defined as Polymorphonuclear count > 250 in ascitic fluid.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No